CLINICAL TRIAL: NCT01410916
Title: An Open-Label, Multi-Center Trial of Eculizumab in Patients With Shiga-Toxin Producing Escherichia Coli Hemolytic-Uremic Syndrome (STEC-HUS)
Brief Title: Safety and Efficacy Study of Eculizumab in Shiga-Toxin Producing Escherichia Coli Hemolytic-Uremic Syndrome (STEC-HUS)
Acronym: STEC-HUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C11-001; 2011-002691-17 (EudraCT Number)
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Shiga-like Toxin-producing Escherichia Coli
Keywords: STEC-HUS; Shiga-like toxin-producing Escherichia Coli Hemolytic-Uremic Syndrome; uncontrolled complement activation
MeSH Terms: interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Eculizumab (Soliris®) — Eculizumab 300 mg, 600 mg, 900 mg or 1200 mg will be administered intravenously

SUMMARY:
This protocol is designed to collect safety and efficacy data on patients that have been or will be treated with eculizumab for STEC-HUS, in the context of the 2011 STEC-HUS epidemic in Germany.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be willing and able to give written informed consent/Assent.
2. Adults, adolescents, or pediatric (≥2 months and ≥5kg) patients
3. Patient has been diagnosed with Escherichia Coli Hemolytic-Uremic Syndrome (STEC-HUS)

Exclusion Criteria:

1. Known complement regulatory mutation or family history of complement regulatory mutation
2. Unresolved systemic meningococcal disease
3. 3. Hypersensitivity to eculizumab, to murine proteins or to one of the excipients

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Improvement in Systemic TMA & Vital Organ Involvement at 8 weeks of treatment defined as either complete or partial responder based on hematologic normalization/improvement & clinically important improvement in Vital Organs: Brain, Kidney, and Thrombosis | 8 weeks
  Analysis of primary endpoint will occur after all patients have reached 8 weeks of treatment. The response rate will be summarized as patients who are either a complete or partial responder.

CONTACTS AND LOCATIONS:
Locations (19):
- Germany (19):
  - Bielefeld
  - Bonn
  - Bremen
  - Bremerhaven
  - Cologne
  - Essen
  - Flensburg
  - Göttingen
  - Hamburg
  - Hanover
  - Karlsruhe
  - Lübeck
  - Magdeburg
  - Munich
  - München
  - Münster
  - Oldenburg
  - Ulm
  - Wildeshausen